CLINICAL TRIAL: NCT02776917
Title: A Phase 1b Pilot Clinical Trial of Cirmtuzumab, an Anti-ROR1 Monoclonal Antibody, in Combination With Paclitaxel for the Treatment of Patients With Metastatic, or Locally Advanced, Unresectable Breast Cancer
Brief Title: Study of Cirmtuzumab and Paclitaxel for Metastatic or Locally Advanced, Unresectable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Parker, MD (Other)
Collaborators: Oncternal Therapeutics, Inc (Industry)
Responsible Party: Sponsor-Investigator, Barbara Parker, MD, Clinical Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160178
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasms
Keywords: metastatic breast cancer; locally advanced, unresectable breast cancer; HER2/NEU negative
MeSH Terms: conditions — Breast Neoplasms | interventions — cirmtuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cirmtuzumab + Paclitaxel (Experimental): Cirmtuzumab 600 mg is administered intravenously on Days 1 and 15 of the first 28-day cycle, then on Day 1 of each subsequent 28-day cycle.
  Paclitaxel 80 mg/m^2 is administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: Cirmtuzumab + Paclitaxel

INTERVENTIONS:
Drug: Cirmtuzumab + Paclitaxel — Cirmtuzumab and paclitaxel may be administered until disease progression or unacceptable toxicity. Cirmtuzumab or paclitaxel may be continued alone if the other drug is discontinued due to toxicity.
  Other Names: UC-961 or Zilovertamab; Taxol

SUMMARY:
This is a pilot phase 1b study to investigate the safety and side effects of combining the ROR1-targeting monoclonal antibody, cirmtuzumab, with paclitaxel for patients with HER2 negative, metastatic breast cancer. Cirmtuzumab is a type of drug called a monoclonal antibody. This drug is designed to attach to a protein called receptor-tyrosine-kinase like orphan receptor 1 (ROR1) on the surface of breast cancer cells. Cirmtuzumab blocks the growth and survival of the breast cancer cells in laboratory tests. ROR1 is rarely expressed on healthy cells. Cirmtuzumab is considered experimental and is not approved by United States (U.S.) Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
* This is a phase 1b, open-label, non-randomized, fixed dose study in patients with HER2 negative metastatic, or locally advanced, unresectable breast cancer.
* Cirmtuzumab and paclitaxel will be administered until disease progression or unacceptable toxicity. Cirmtuzumab or paclitaxel may be continued alone if the other drug is discontinued due to toxicity, as long as the subject is tolerating the drug and does not exhibit disease progression.
* Blood and tissue samples will be collected at pre-specified times to enable pharmacokinetic and correlative studies.
* Adverse events (AE) will be monitored throughout the trial. Reporting of AEs will be in accordance with CTCAE version 4.03.
* Assessment of tumor response will be performed by physical examination and/or by radiographic imaging and according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
* Patients will be assessed at 28 days following the last dose of cirmtuzumab to assess tumor response and at 56 days following the last dose of cirmtuzumab to assess any adverse events and to document any concomitant cancer therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

* Biopsy-confirmed, metastatic or locally advanced surgically unresectable, HER2 negative breast cancer. HER2 status should reflect the most recent biopsy results. Note: HER2 negative breast cancer is defined according to the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines 2013 for HER2 testing performed in a CLIA-certified laboratory.
* ER/PR negative (<10% of cells staining for ER or PR) breast cancer or have ER/PR positive (≥10% of cells staining for ER or PR) breast cancer that has exhausted standard endocrine therapy and/or in the opinion of the treating oncologist, warrants cytotoxic chemotherapy.
* Measurable disease as defined by RECIST v1.1. Measurable lesions will be confirmed by radiographic imaging (CT or MRI). Patients with bone only disease will be eligible if disease is considered measurable and a soft tissue component is present and can be biopsied..
* There is no limit to prior lines of therapy, but patients must not have received prior taxane chemotherapy in the metastatic setting.
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined below:

  * Absolute Neutrophil Count ≥ 1.0 x 10^9/L
  * Platelet count ≥ 100,000 /μL
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal
  * AST and ALT ≤ 3 x upper limit of normal
  * Serum creatinine ≤ 2 x upper limit of normal OR Creatinine clearance > 40 ml/min/1.73 m^2
* Women of child-bearing potential and male subjects who are sexually active with a woman of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months following last infusion of cirmtuzumab. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Existing neuropathy must be no greater than Grade 1.
* No concurrent antibody therapy can be planned with the exception of denosumab for use in bone metastasis.
* CNS metastases are allowed as long as the metastases are asymptomatic, have been treated with radiation, and have been stable for > 6 weeks off steroids.

EXCLUSION CRITERIA:

* Patient is currently receiving chemotherapy or has received another chemotherapy within 5 half-lives, radiotherapy or immunotherapy within 2 weeks prior to study treatment initiation.
* Patient has known, untreated and/or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Patient had disease that was refractory to paclitaxel in the neoadjuvant setting and/or developed metastatic breast cancer within 6 months of neoadjuvant or adjuvant taxane chemotherapy.
* Patient has had major surgery within 3 weeks prior to enrollment.
* Patient has severe and/or uncontrolled medical disease(s) (i.e., myocardial infarction within 6 months of study, CKD stage IV or above, severe chronic pulmonary disease or active infection).
* The patient has known acute or chronic hepatitis B or C.
* The patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel.
* The patient has a history of another malignancy within 2 years prior to study entry, except curatively treated non-melanotic skin cancer, cervical carcinoma in situ or stage I colon cancer.
* Patient has a history of non-compliance or other medical illness that would preclude compliance with study procedures.
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient has severe cardiac insufficiency (NYHA III or IV) with uncontrolled and/or unstable cardiac or coronary artery disease
* Patient is pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Parker, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shatsky RA, Batra-Sharma H, Helsten T, Schwab RB, Pittman EI, Pu M, Weihe E, Ghia EM, Rassenti LZ, Molinolo A, Cabrera B, Breitmeyer JB, Widhopf GF 2nd, Messer K, Jamieson C, Kipps TJ, Parker BA. A phase 1b study of zilovertamab in combination with paclitaxel for locally advanced/unresectable or metastatic Her2-negative breast cancer. Breast Cancer Res. 2024 Feb 26;26(1):32. doi: 10.1186/s13058-024-01782-0. PMID 38408999
- See also: PubMed — https://pubmed.ncbi.nlm.nih.gov/38408999/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cirmtuzumab + Paclitaxel: Cirmtuzumab 600 mg is administered intravenously on Days 1 and 15 of the first 28-day cycle, then on Day 1 of each subsequent 28-day cycle.
  Paclitaxel 80 mg/m^2 is administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle.
  Cirmtuzumab + Paclitaxel: Cirmtuzumab and paclitaxel may be administered until disease progression or unacceptable toxicity. Cirmtuzumab or paclitaxel may be continued alone if the other drug is discontinued due to toxicity.
Period: Overall Study
Arm/Group | Cirmtuzumab + Paclitaxel
Started | 23
Completed | 16
Not Completed | 7
Not completed — Screen failures. One subject ended treatment early due to disease related symptoms | 7

BASELINE CHARACTERISTICS:
Population: Participants who completed at least 4 weeks of treatment
Arm/Group | Cirmtuzumab + Paclitaxel
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.56 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities During the First 4 Weeks of Treatment
Description: Clinically significant adverse events per CTCAE Version 4.03 at least possibly related to cirmtuzumab or the combination of cirmtuzumab and paclitaxel during the first four weeks of investigational treatment.
Time Frame: Within 4 weeks of starting study treatment
Measure: Number; unit: participants
Arm/Group | Cirmtuzumab + Paclitaxel
Number analyzed (Participants) | 16
participants | 0

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events beginning from the start of study treatment to 30 days after study treatment completion or start of new anti-cancer therapy.
Time Frame: 55 weeks
Measure: Number; unit: participants
Arm/Group | Cirmtuzumab + Paclitaxel
Number analyzed (Participants) | 16
participants | 16

3. Secondary Outcome: Objective Tumor Response Rate
Description: Response and progression were evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines.
Time Frame: 55 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cirmtuzumab + Paclitaxel
Number analyzed (Participants) | 16
Participants | 6

4. Secondary Outcome: Best Tumor Response Rate
Description: The proportion of patients that achieve a response of stable disease or better as assessed by RECIST v1.1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cirmtuzumab + Paclitaxel
Number analyzed (Participants) | 16
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse events were monitored weekly from the beginning of study procedures to 30 days following the last administration of study treatment or start of new anti-cancer therapy. The median time on study was 16 weeks with a median number of cycles ranging from 1 to 14.
Arm/Group | Cirmtuzumab + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirmtuzumab + Paclitaxel (N=16)
Back Pain (General disorders) | 1 (1) — Grade 3 Adverse Event. Not Related to Taxol attribution and Not Related to Cirmtuzumab attribution
Joint range of motion decreased cervical spine (General disorders) | 1 (1) — Grade 3 Adverse Event. Not Related to Taxol attribution and Not Related to Cirmtuzumab attribution
Flu like symptoms (Immune system disorders) | 1 (1) — Grade 3 Adverse Event. Probably related to Taxol attribution and Unlikely related to Cirmtuzumab attribution
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Grade 3 Adverse Event. Not Related to Taxol attribution and Not Related to Cirmtuzumab attribution
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 3 Adverse Event. Not Related to Taxol attribution and Not Related to Cirmtuzumab attribution
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirmtuzumab + Paclitaxel (N=16)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Blurred vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 9 (12)
Diarrhea (Gastrointestinal disorders) | 7 (11)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (14)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 3 (4)
Fatigue (General disorders) | 13 (14)
Fever (General disorders) | 4 (4)
Flu like symptoms (General disorders) | 5 (8)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (4)
Pain (General disorders) | 6 (12)
Infections and infestations - Other, specify (Infections and infestations) | 2 (5)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 6 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (8)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (8)
Urinary retention (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (3)
Flushing (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT02776917/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT02776917/SAP_001.pdf